CLINICAL TRIAL: NCT07172711
Title: Subtype-Specific Catheter-Related Bloodstream Infection Risk Factors in Hospitalized Patients With Intestinal Failure: A Retrospective Study
Brief Title: Risk Factors for Catheter-Related Bloodstream Infections in Hospitalized Intestinal Failure Patients
Status: Completed | Type: Observational
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Wang Xinying, Professor of Medicine, Jinling Hospital, China
Other Study IDs: 20250901
Record Dates: First submitted 2025-09-01; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Catheter-related Bloodstream Infection; Intestinal Failure
MeSH Terms: conditions — Intestinal Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CRBSIs: Patients with intestinal failure who developed catheter-related bloodstream infection
- Non-CRBSI: Patients with intestinal failure who never developed catheter-related bloodstream infection

SUMMARY:
This retrospective cohort study aims to identify risk factors for catheter-related bloodstream infections (CRBSIs) in hospitalized patients with intestinal failure (IF), including all subtypes (Types I-III). The study included 321 patients with 9,365 catheter-days. Multivariate logistic and Cox regression analyses were used to identify independent risk factors. Stratified analyses identified subtype-specific risks, and hospital stay length and health economic outcomes were assessed. The study highlights the need for subtype-tailored prevention strategies and closer metabolic and immune monitoring in hospitalized IF patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the ESPEN 2023 diagnostic criteria for intestinal failure.

Exclusion Criteria:

* Catheter indwelling duration <48 hours; Implanted catheter before admission; Complex components in PN difficult to quantify; Positive blood cultures with unclear CRBSI diagnosis; Alternative infection sources identified.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This single-center retrospective study enrolled 321 patients with intestinal failure admitted between 2021 and 2024. All included patients met the ESPEN 2023 diagnostic criteria for intestinal failure, defined as reduced intestinal function below the minimum necessary for absorption of macronutrients and/or water-electrolytes, thus requiring intravenous supplementation (IVS) to maintain health and/or growth. Patients were excluded if they met any of the following criteria: Catheter indwelling duration <48 hours; Implanted catheter before admission; Complex components in PN difficult to quantify; Positive blood cultures with unclear CRBSI diagnosis; Alternative infection sources identified.
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
incidence rate of catheter-related bloodstream infection | From catheter insertion until removal or discharge, assessed up to 24 months.
  frequency of catheter-related bloodstream infections occurring every 1,000 days

SECONDARY OUTCOMES:
Proportion of patients with high calorie-to-nitrogen ratio | From catheter insertion until removal or discharge, assessed up to 24 months.
  The proportion of patients receiving a parenteral nutrition formula with a non-protein calorie-to-nitrogen ratio (C/N ratio) equal to or greater than 100 kilocalories per gram of nitrogen (≥100 kcal/g N).
Incidence of lymphocytopenia | Baseline.
  The proportion of patients with lymphocytopenia at baseline.
Proportion of patients with high parenteral nutrition energy supply | From catheter insertion until removal or discharge, assessed up to 24 months.
  The proportion of patients whose average proportion of daily energy from PN to measured resting energy expenditure (PN/REE) exceeds 0.6 during the catheter indwelling period.
Incidence of neutropenia | Baseline
  The proportion of patients with neutropenia at baseline.
All-cause length of hospital stay | At the time of hospital discharge, assessed up to 24 months.
  The total duration of hospitalization, measured in days, from admission to discharge.
Total hospitalization costs | At the time of hospital discharge, assessed up to 24 months.
  The total direct medical costs (in CNY) incurred during the hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Wang, Study Chair — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No